CLINICAL TRIAL: NCT00644982
Title: A Multicenter Randomized, Double-Blind, Parallel-Group Study of Sertraline Versus Venlafaxine XR in the Acute Treatment of Outpatients With Major Depressive Disorder
Brief Title: A Comparison of Sertraline Versus Venlafaxine XR in the Treatment of Major Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0501066
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sertaline group (Experimental)
  Interventions: Drug: sertraline
- Venlafaxine group (Active Comparator)
  Interventions: Drug: venlafaxine XR

INTERVENTIONS:
Drug: sertraline — Flexibly-titrated 50 mg tablets, 50-150 mg/day and venlafaxine placebo orally for 10 weeks.
  Other Names: Zoloft
  Arms: Sertaline group
Drug: venlafaxine XR — Flexibly-titrated 75 mg capsules, 75-225mg/day and sertraline placebo orally for 10 weeks.
  Arms: Venlafaxine group

SUMMARY:
To assess the comparative efficacy of sertraline versus venlafaxine XR on measures of quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of DSM-IV Major Depressive Disorder, single episode or recurrent, without psychotic features. Additional DSM-IV Axis I diagnoses will be permitted only if they are identified as secondary diagnoses.
* Hamilton-Depression rating scale (HAM-D; 17 item) total score ≥18 and HAMD item 1 (depressed mood) score ≥2.

Exclusion Criteria:

* Use of an antidepressant within 2 weeks of baseline (4 weeks for fluoxetine)
* Current or past diagnosis of bipolar disorder or any psychotic disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2002-10; Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QOL, measured using the Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q). | Weeks 1, 2, 3, 4, 6, 8, 9 and 10.

SECONDARY OUTCOMES:
Change from baseline in the 17-item Hamilton-Depression Rating Scale (HAM-D) including response (≥50% reduction in HAM-D total score from baseline) and remission (HAM-D total score ≤7) rates. | Weeks 1, 2, 3, 4, 6, 8, 9 and 10.
The 17-item Hamilton-Depression Rating Scale response rates at endpoint (week 8). | Week 8
CGI response rate at endpoint (week 8). | Week 8
Change from baseline in the CGI-Severity Scale (CGI-S). | Weeks 1, 2, 3, 4, 6, 8, 9 and 10.
Change from baseline in the Hamilton Anxiety Scale (HAM-A). | Weeks 1, 2, 3, 4, 6, 8, 9 and 10.
Change from baseline in the Endicott Work Productivity Scale (EWPS). | Weeks 1, 8, 9, 10
Change from baseline in the Visual Analogue Scale (VAS) for Depression. | Weeks 1, 2, 3, 4, 6, 8, 9 and 10.
Change from baseline in the Visual Analogue Scale (VAS) for Overall Assessment of Pain. | Weeks 1, 2, 3, 4, 6, 8, 9 and 10.
Hamilton-Depression Rating Scale remission rates at endpoint (week 8). | Week 8
Change from baseline in the Clinical Global Impression-Improvement Scale. | Weeks 1, 2, 3, 4, 6, 8

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- Australia (7):
  - Pfizer Investigational Site, Cairns, Queensland
  - Pfizer Investigational Site, Everton Park, Queensland
  - Pfizer Investigational Site, North Cairns, Queensland
  - Pfizer Investigational Site, Box Hill, Victoria
  - Pfizer Investigational Site, Heidelberg, Victoria
  - Pfizer Investigational Site, WEST Heidelberg, Victoria
  - Pfizer Investigational Site, West Perth, Western Australia
- Turkey (Türkiye) (7):
  - Pfizer Investigational Site, Adana
  - Pfizer Investigational Site, Ankara
  - Pfizer Investigational Site, Diyarbakır
  - Pfizer Investigational Site, Istanbul
  - Pfizer Investigational Site, Izmir
  - Pfizer Investigational Site, İzmit
  - Pfizer Investigational Site, Malatya

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0501066&StudyName=A%20comparison%20of%20Sertraline%20versus%20Venlafaxine%20XR%20in%20the%20treatment%20of%20major%20depression.